CLINICAL TRIAL: NCT06811480
Title: The Effectiveness of Closed Kinetic Chain Exercises in Individuals With a Distal Radius Fracture
Brief Title: Effectiveness of Closed Kinetic Chain Exercises in Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: burak menek (Other)
Responsible Party: Sponsor-Investigator, burak menek, Principal Investigator, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-10840098-202.3.02-7483
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Distal Radius Fractures
Keywords: Closed kinetic chain exercises (CKCE); Rehabilitation; Proprioception; Distal Radius Fractures
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional physiotherapy (CP) group (Active Comparator): Participants in the first group underwent conventional physiotherapy interventions for 6 weeks, 5 days per week.
  Interventions: Other: Conventional Physiotherapy
- closed kinetic chain exercises (CKCE) group (Experimental): Participants in the second group received a treatment protocol including closed kinetic chain exercises (CKCE) in addition to conventional physiotherapy interventions.
  Interventions: Other: Conventional Physiotherapy; Other: Closed Kinetic Chain Exercise

INTERVENTIONS:
Other: Conventional Physiotherapy — Participants in the first group underwent conventional physiotherapy interventions for 6 weeks, 5 days per week. These interventions included Ultrasound (US), Transcutaneous Electrical Nerve Stimulation (TENS), wrist joint range of motion exercises, stretching exercises, and strengthening exercises using Digiflex, Powerweb, and dumbbells. The number of repetitions and sets of the exercises was adjusted based on the patients' conditions, following a progressive approach.
  US was applied to the affected wrist for a total of 30 sessions, 5 days a week, once daily, for 6 minutes at an intensity of 1.5 W/cm², using an underwater application method. TENS was administered at a frequency of 100 Hertz for 20 minutes. All participants received manual stretching exercises for wrist flexion, extension, ulnar and radial deviation, supination, and pronation. These stretches were performed by a physiotherapist, with 5 repetitions in each direction, holding the end position for 20 seconds.
Other: Closed Kinetic Chain Exercise — Participants in the second group received a treatment protocol that included closed kinetic chain exercises (CKCE) in addition to conventional physiotherapy. CKCE exercises were performed with 15 repetitions each and involved stabilizing a ball between the hand and the wall in different arm positions, rolling it in multiple directions. Participants also performed weight-shifting exercises against a wall and on a table, holding positions for 6 seconds. Additionally, in a crawling position, they moved their unaffected arm diagonally on both a firm surface and a cushion.
  Arms: closed kinetic chain exercises (CKCE) group

SUMMARY:
The aim of this study is to evaluate the effectiveness of closed kinetic chain exercises during the physiotherapy and rehabilitation process following the healing of a distal radius fracture.

A total of 40 participants aged 40-60 years who were diagnosed with distal radius fractures were randomly assigned to two groups: the conventional physiotherapy (CP) group (n=20) and the closed kinetic chain exercise (CKCE) group (n=20). Participants in the CP group underwent a 6-week standard rehabilitation program consisting of conventional physiotherapy sessions conducted 5 days a week. This program included Ultrasound (US), Transcutaneous Electrical Nerve Stimulation (TENS), wrist joint range of motion exercises, stretching exercises, Digiflex, Powerweb, and dumbbell-based strengthening exercises. In the CKCE group, the same CP program was implemented with the addition of CKCE sessions conducted five days a week for 6 weeks.

Outcome measures included joint range of motion assessed using the Goniometer Pro mobile application, functionality evaluated with the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, pain intensity measured using the Visual Analog Scale (VAS), and joint position sense assessed through the Active Repositioning Test.

CKCE may positively affect joint range of motion, arm functionality, pain, and joint position sense by improving the proprioceptive mechanism in individuals with distal radius fractures.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effectiveness of closed kinetic chain exercises during the physiotherapy and rehabilitation process following the healing of a distal radius fracture.

Voluntary consent forms were signed by individuals willing to participate in the study, and their demographic information was recorded. A total of 40 participants were included in the study and divided into two groups:

Group 1: Conventional Physiotherapy Group (n=20) Group 2: Closed Kinetic Chain Exercise Group (n=20) Participants in the first group underwent conventional physiotherapy interventions for 6 weeks, 5 days per week. These interventions included Ultrasound (US), Transcutaneous Electrical Nerve Stimulation (TENS), wrist joint range of motion exercises, stretching exercises, and strengthening exercises using Digiflex, Powerweb, and dumbbells. The number of repetitions and sets of the exercises was adjusted based on the patients' conditions, following a progressive approach.

US was applied to the affected wrist for a total of 30 sessions, 5 days a week, once daily, for 6 minutes at an intensity of 1.5 W/cm², using an underwater application method. TENS was administered at a frequency of 100 Hertz for 20 minutes. All participants received manual stretching exercises for wrist flexion, extension, ulnar and radial deviation, supination, and pronation. These stretches were performed by a physiotherapist, with 5 repetitions in each direction, holding the end position for 20 seconds.

Participants in the second group received a treatment protocol including closed kinetic chain exercises (CKCE) in addition to conventional physiotherapy interventions. As part of the CKCE program, the following exercises were performed with 15 repetitions each:

While the elbow was in extension and the shoulder was at 90° flexion, a ball was stabilized between the hand and the wall. The ball was rolled up and down as well as side-to-side.

While the elbow was in extension and the shoulder was at 90° abduction, a ball was stabilized between the hand and the wall. The ball was rolled up and down as well as side-to-side.

While the elbow was in extension and the shoulder was at 90° flexion, participants were asked to push against the wall by transferring body weight from the shoulder to the elbow and wrist. They held this position for 6 seconds.

Randomization:

The study included 40 participants aged between 40-60 years who were diagnosed with distal radius fractures. A computer-based randomization program was used to assign participants to groups. The randomization codes were sealed in envelopes, which were opened by the physiotherapist administering the exercises on the day of the intervention.

Outcome Measures:

Outcome measures included joint range of motion assessed using the Goniometer Pro mobile application, functionality evaluated with the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, pain intensity measured using the Visual Analog Scale (VAS), and joint position sense assessed through the Active Repositioning Test.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 40-60 years
* Diagnosed with a distal radius fracture
* Applied to Medipol hospitals after the injury and volunteered to participate in the study
* Patients with good cooperation levels will be included in the study

Exclusion Criteria:

* Having bilateral distal radius fractures
* Having ulna styloid fractures
* Having other orthopedic, neurological, or rheumatological problems involving the ipsilateral upper extremity
* A history of surgery involving the ipsilateral upper extremity
* Associated injuries such as arterial, nerve, or tendon injuries
* Patients without adequate cooperation will be excluded from the study

Withdrawal Criteria:

* Missing at least one follow-up
* Development of orthopedic or systemic problems unrelated to the trauma

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-06 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
JPS testing | From enrollment to the end of treatment at 8 weeks
  Joint position sense (JPS) testing was conducted using a standardized protocol with a goniometer for active wrist position measurement. Participants, seated with their elbow flexed on a table, had their wrist passively moved to 30º extension to memorize the position. With vision occluded, they moved their wrist to full flexion and attempted to reproduce the 30º extension. The reproduced wrist position was recorded, and the difference from the reference angle determined the JPS deficit. A zero value indicated perfect reproduction, while absolute differences reflected the deficit's magnitude. Two trials' mean values were used for analysis.
Goniometric Measurement | From enrollment to the end of treatment at 8 weeks
  In this study, the affected shoulder's flexion, extension, abduction, internal rotation, and external rotation angles will be measured using a goniometer-pro application. Reference values will include 0-180 degrees for flexion and abduction, 45 degrees for extension, and 0-90 degrees for internal and external rotation

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | From enrollment to the end of treatment at 8 weeks
  The Visual Analog Scale (VAS) is a commonly used tool in clinical settings for assessing pain intensity. Participants rate their pain on a scale from 0 to 10, where 0 indicates no pain, and 10 represents unbearable pain. Pain intensity at rest and during activity will be evaluated using the VAS for participants before and after the treatment
Disabilities of the Arm, Shoulder, and Hand (DASH) | From enrollment to the end of treatment at 8 weeks
  The DASH questionnaire, introduced in collaboration with the American Academy of Orthopedic Surgeons and other organizations, evaluates physical limitations and functionality in upper extremity problems (10). The DASH consists of three subsections. The first section includes 30 questions: 21 assess difficulties in daily living activities, 5 evaluate symptoms, and 4 measure social function, work, sleep, and self-confidence. An optional module (Work Module (DASH-W)) with 4 additional questions assesses the impact on work life

CONTACTS AND LOCATIONS:
Locations (1):
- Burak Menek, Istanbul, Beykoz, Turkey (Türkiye)

REFERENCES:
- [Derived] Menek B, Dansuk E. Investigating the effects of closed kinetic chain exercises on joint position sense, functionality, range of motion, and pain in individuals with distal radius fracture: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2025 May 31;17(1):137. doi: 10.1186/s13102-025-01195-2. PMID 40450369